CLINICAL TRIAL: NCT03430570
Title: An Emotion Regulation Intervention for Early Adolescent Risk Behavior Prevention
Brief Title: An Emotion Regulation Intervention for Early Adolescent Risk Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21HD089979 (NIH); R21HD089979 (NIH)
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-02

CONDITIONS: Risk Behavior; Risk Reduction; Emotion Regulation
Keywords: Adolescent risk behavior; digital; early adolescence; emotion regulation; prevention
MeSH Terms: conditions — Risk-Taking; Risk Reduction Behavior; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to complete a computerized intervention or a wait list control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tablet TRAC Emotion Regulation Intervention (Experimental)
  Interventions: Behavioral: Tablet TRAC Emotion Regulation Intervention
- Waitlist Control (No Intervention): Control participants are assessed on the same schedule as the treatment condition and offered the intervention after the 3-month follow-up

INTERVENTIONS:
Behavioral: Tablet TRAC Emotion Regulation Intervention — The intervention focuses on developmentally appropriate strategies for emotion regulation during difficult situations, particularly those related to risk, using 3 primary groups of strategies identified during qualitative work in Project TRAC (R34 MH078750): 1) getting away (physically or cognitively) from triggers for strong emotions, 2) releasing emotional energy in healthy ways (physically or verbally) or 3) changing cognitions and appraisals about emotional triggers. Using strategies effective in TRAC, teens will engage in games to practice and apply strategies to risk scenarios, as well as personalize content learned.
  Arms: Tablet TRAC Emotion Regulation Intervention

SUMMARY:
This study will take a group-based intervention for adolescents that reduced sexual risk behavior and create a computer-based version, which is a format that adolescents like and that is more cost-effective. The intervention focuses on teaching adolescents skills for managing their emotions when they are making decisions that could put them at risk (like whether to have sex or drink alcohol). The investigators are hoping to learn whether a computer version of the program will be useful in helping adolescents learn about emotional competence and reducing risky behaviors. The investigators will make a version of the intervention as games on tablet computers in a partnership with a technology company, Klein Buendel. The research team will begin by getting advice from adolescents and experts (in separate groups) about how to convey the ideas from the group program into computer games. Klein Buendel will then create the games. Then, about 10 adolescents will be asked to try out the program and give us feedback about things to change. Klein Buendel will make those changes. Then the investigators will ask about 100 adolescents to volunteer to be randomly placed in one of two groups. One group will do the computer program right away; the other will wait for three months. Both groups will be asked to answer questions and do computer tasks when the team meets them, one month later, and three months later. The investigators will compare the groups to see if the group that received the computer intervention reports being more emotionally competent than the group that has not yet done the computer intervention. The research team will also ask them about their risk behaviors. If this is useful, it may be a good way to enhance health education taught in schools.

DETAILED DESCRIPTION:
Emotion regulation in adolescence is associated with health risk behaviors, including sex and substance use, and early onset of these behaviors represents a risk factor for negative health outcomes throughout life. Thus, interventions appropriate for early adolescence, when these behaviors commonly begin, are critical for prevention efforts. The research team has developed and tested a novel, engaging, and efficacious intervention that addresses emotion regulation, a theoretically important and under-researched factor associated with risk. The efficacy trial of this intervention, Project TRAC, showed that an intervention strategy using emotion regulation was significantly more successful than an active comparison condition on the primary target, delaying onset of sexual activity over a two and a half year follow-up, as well as on other risk behaviors, such as condom use, fighting, and partner violence. While efficacious, the current face-to-face, small group format of the program is a difficult model to sustain and implement on a larger scale. With a long-term goal toward dissemination, this two-year project will translate the emotion regulation components of this successful program for tablet-based delivery to enable it to reach a large audience in a format that can be related to a variety of health behavior education topics (e.g., sexual health, violence, substance use). For the proposed project, the Rhode Island Hospital/ Brown University research team will collaborate with Klein Buendel, a health communications technology company, to translate the emotion regulation content of Project TRAC for tablet computers. This translation, using well-established theoretical frameworks, will be approached in consultation with members of the target population (early adolescents) and experts in the field. After the intervention has been translated to a tablet form, ten adolescents will test the program to assess acceptability and usability. Finally, a small pilot study (n=100) will assess feasibility of the translated intervention and compare it to a waitlist control group.

ELIGIBILITY:
Inclusion Criteria:

* attending the seventh grade at a participating school
* being between the ages of 12 and 14

Exclusion Criteria:

* those who cannot read English at a 4th grade level
* those with developmental delays

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Emotion Regulation/Difficulties in Emotion Regulation Scale | baseline- 3 month follow up
  Difficulties in Emotion Regulation Scale- The Difficulties in Emotion Regulation Scale (36 items) uses 6 subscales (all α > .80) to assess perceptions of skill in ER, awareness, and impulse control based on Linehan's theoretical work.
  The six subscales are:
  1. Nonacceptance of emotional response (6 items)
  2. Difficulties engaging in goal directed behavior [goals] (5 items)
  3. Impulse control difficulties [impulse] (6 items)
  4. Lack of emotion awareness [awareness] (6 items)
  5. Limited access to emotion regulation strategies [strategies] (8 items)
  6. Lack of emotional clarity [clarity]. (5 items)
  Participants rate their responses on a 5-point Likert scale ranging from 1 (almost never)- 5 (almost always). The total score is calculated from the sum of all the items, with higher scores indicating greater problems with emotion regulation. (Total possible range: 36-180)

SECONDARY OUTCOMES:
Emotion Recognition/DANVA | Baseline-3 month follow up
  Diagnostic Analysis of Nonverbal Accuracy-2 (DANVA2) is a computer-based measure that asks participants to identify the emotion of facial expressions displayed in a series of 24 photographs and in 24 oral presentations of a neutral sentence, with higher scores indicating higher accuracy of emotion recognition. Total possible range = 0-48.
Emotion Regulation/Emotion Regulation Checklist | baseline-3 month follow up
  The Emotion Regulation Checklist contains 24 items on a 4-point Likert scale (1=never through 4= almost always; Total Range: 15-360). Parents rate 24 behavioral descriptions, yielding 2 subscales: 1) Lability/Negativity (α= .95), and 2) Emotion Regulation (α=.84). The Emotion Regulation subscale contains 8 items, while the Lability/Negativity scale contains 15 items. Higher scores on the Lability/Negativity scale indicate higher inflexibility, emotional reactivity, and dysregulated negative affect; higher scores on the emotion regulation subscale indicate greater situationally appropriate affective displays, empathy, and emotional self-awareness (Shields & Cicchetti, 1997). Alphas for the subscales are good (L/N α = .96; ER α = .83). One single measurement of emotion regulation is generated from the overall scores in both sub-scales (α = .89; Shields & Cicchetti, 1997).
Emotion Regulation/ The Regulation of Emotions Questionnaire | baseline-3 month follow up
  The Regulation of Emotions Questionnaire* (21 items) assesses frequency of use of both functional and dysfunctional emotion regulation strategies (α= >.66). Participants rate their responses on a 5-point Likert scale from 1- "never" through 5- "always". (Total Range: 21-110). Higher scores indicate higher frequency of use of emotion regulation strategies.
Emotion Regulation/Self Efficacy Questionnaire for Children | baseline-3 month follow-up
  The Emotional Self-efficacy subscale of the Self-Efficacy Questionnaire for Children (8 items) assesses perception of one's ability to cope with negative emotions (α= .83). It has been shown to be valid, reliable, and related to risk behaviors among US adolescents. Subjects rate their responses on a 5-point Likert scale from 1 "not at all" through 5 "very well". (Range: 8-40, with lower scores indicating low perception of ability to cope with negative emotions).
Emotion Regulation/Emotion Regulation Behavior Scale | baseline-3 month follow up
  The Emotion Regulation Behaviors Scale (8 items) measures use of the specific emotion regulation strategies taught in Project TRAC (α= .73). Participants respond on a scale of 1 (never) to 5 (all the time) across 8 items, with higher scores indicating more regulatory behaviors (range: 8-40).
Emotion Regulation/Affect Dysregulation Scale | baseline-3 month follow up
  The Affect Dysregulation Scale contains 6 items used to assess frequency of difficulty with affect regulation on 4-point Likert scale from 1=not at all to 4=often (α= .72), with higher scores indicating more difficulty managing feelings. affect (range: 6-36).
Assessment Risk Behavior/Youth Risk Behavior Surveillance System | Baseline-3 month follow up
  7 items taken from the Center for Disease Control's Youth Risk Behavior Surveillance System will be used to assess adolescents' engagement in substance use, violence, and other risk behaviors. Participants will be asked risk behavior questions similar to the following item: "During the past 30 days, on how many days did you smoke cigarettes?" with answer choices ranging from 0, 1-2, 3-5, 6-9, 10-19, 20-29, 30.
Distress Tolerance | baseline-3 month follow up
  Behavioral Indicator of Resiliency to Distress (BIRD) and Mirror Tracing Persistence Task (MTPT) are 5-minute computerized distress tolerance tasks that generate a score of time spent persisting on a dysregulating task that provides negative feedback (aversive noise) when users do not succeed at very challenging tasks, with more time spent on the tasks indicating greater distress tolerance. Possible range = 0-300 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Houck, PhD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital- Bradley Hasbro Children's Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
After analyses are completed for the aims of the study, deidentified databases will be made available to qualified researchers through standard data sharing procedures.